CLINICAL TRIAL: NCT06641271
Title: Vagus Nerve Stimulation to Promote Remyelination in Multiple Sclerosis
Brief Title: Study to Investigate Vagus Nerve Stimulation Paired With Motor Task for Remyelination and Functional Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-1451
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental - Active Stimulation (Experimental): Participants in this arm will receive active stimulation during the paired motor task.
  Interventions: Device: Closed Loop Trans-Auricular Vagus Nerve Stimulation System
- Control - Sham Stimulation (Sham Comparator): Participants in this arm will receive sham stimulation during the paired motor task to create a control to the experimental group.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Closed Loop Trans-Auricular Vagus Nerve Stimulation System — A closed loop system that delivers stimulation to the vagus nerve via the ear non-invasively following a trigger event.
  Arms: Experimental - Active Stimulation
Device: Placebo — A closed-loop vagus nerve stimulation device that can deliver sham stimulation to the ear to simulate stimulation of the vagus nerve.
  Arms: Control - Sham Stimulation

SUMMARY:
The goal of this clinical trial is to learn if stimulating the vagus nerve in combination with a motor task in people with multiple sclerosis can improve motor function. The main questions it aims to answer are:

* Is stimulating the vagus nerve safe and feasible after demyelinating episodes?
* Does a paired motor task with vagus nerve stimulation improve motor function with someone who has multiple sclerosis?

Researchers will compare active vagus nerve stimulation to a sham stimulation to see if the paired vagus nerve stimulation can improve motor control.

Participants will:

* Come in for study visits over a six month period. Study visits are three times weekly for the first month, then single follow up visits at two, three, and six months.
* During study visits, participants will complete 30 minutes of the paired vagus nerve stimulation with a motor task, specifically the grooved peg test.
* At various timepoints in the study, motor and disability tests will be administered to see if there are any changes in motor control for that participants. These tests include the timed 25 foot walk test, expanded disability scale, the upper extremity portion of the Fugl-Meyer Assessment, and the Multiple Sclerosis Impact Scale - 29.

ELIGIBILITY:
Inclusion Criteria:

* All participants ages 18-65 with diagnosis of multiple sclerosis at least 30 days from last relapse
* Baseline grooved peg test time greater than or equal to 108 seconds for completion of the task (1 standard deviation below mean multiple sclerosis score).
* Ability to sign informed consent
* expanded disability status scale score (or estimated) of 2.5 or greater OR a clinical report of upper extremity dysfunction in their dominant hand

Exclusion Criteria:

* Current uncontrolled and/or clinically significant medical condition.
* Primary progressive multiple sclerosis.
* History of seizures or epilepsy.
* Other central nervous system disease or significant brain trauma.
* Bacterial or viral infection within the prior 30 days.
* Prior treatment with total body irradiation, clemastine, bexarotene, or other experimental remyelinating agent.
* Recent suicide attempt or continued expressed suicidal ideation.
* Implanted devices, such as pacemakers, cochlear prosthesis, neuro-stimulators.
* Abnormal ear anatomy or ear infection.
* Pregnancy, lactation, or lack of use of contraception.
* Unable to walk 25 feet continuously
* Other significant disease or disorder that might impair study participation. Participants will be allowed to initiate or maintain background disease modifying therapy to reduce the risk of multiple sclerosis relapse and optimize recruitment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in time to complete the grooved peg test | End of Study (6 months)
  The participant will complete the grooved peg test with their dominant hand and will be timed while doing so. The change in time to completion will be tracked over the study.
Change from baseline of score of the upper extremity portion of the Fugl-Meyer Assessment | End of Study (6 months)
  The upper extremity portion of the Fugl-Meyer assessment evaluates movements of the upper limbs with score ranging from 0 - 66. A higher score indicates more function.
Change from baseline score of the Expanded Disability Status Scale | End of Study (6 months)
  The expanded disability status scale scores range from 0 - 10, where 10 indicates full function.
Change in time from baseline to complete the timed 25 foot walk test | End of Study (6 months)
  The timed 25 foot walk test is a performance measure where the participants walks 25 feet unassisted and the time to completion is recorded.
Change from baseline in composite disability metric | End of Study (6 months)
  The fraction of participants in each intervention group at 6 months with improvement in disability will be determined by a composite disability metric composed of three elements: expanded disability status scale, timed 25 foot walk, and grooved peg test time. The metric will be deemed positive if there is a significant change in one or more of the measures as determined as follows: 1) decrease in expanded disability status scale score of 1 point (baseline expanded disability status scale score ≤5.5) or 0.5 point (baseline expanded disability status scale score of >5.5); 2) 20% decrease in timed 25 foot walk test; or 3) 25% decrease in grooved peg test time. The composite disability metric will be quantified by a trained study personnel.
Change from baseline in patient reported outcomes from the multiple sclerosis impact scale 29 | End of Study (6 months)
  The Multiple Sclerosis Impact Scale - 29 is a 29-item patient-reported measure of the physical and psychological impacts of multiple sclerosis. Participants are asked to rate how much their functioning and well-being has been impacted over the past 14 days on a 4-point scale. Higher scores indicate a greater disease impact.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bennett, MD, Principal Investigator — Anschutz Campus - School of Medicine - Neurology
Locations (1):
- Clinical Translational Research Center at CU Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No